CLINICAL TRIAL: NCT01426243
Title: The Yellow Fever Vaccine Immunity in HIV Infected Patients : Development of New Assays for Virological and Immunological Monitoring in HIV Infected Patient
Acronym: EP46 NOVAA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-014921-17
Record Dates: First submitted 2011-02-10; First posted 2011-08-31 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2018-02

CONDITIONS: HIV Infection; Yellow Fever
MeSH Terms: conditions — HIV Infections; Yellow Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voluntary HIV positive subjects (Active Comparator): 40 HIV positive adults under HAART for at least one year (and stable on treatment for at least 3 months prior to enrolment), > 350 CD4/mm3 (with half of them a nadir < 200 CD4/mm3) and a viral load < 50 copies/mL for at least 6 months. Patients were HCV negative or non-replicative and treated for at least 2 years with normal ALT and negative HBs antigen.
  Interventions: Biological: Yellow fever vaccination (STAMARIL)
- HIV negative subjects (Other): Voluntary HIV negative subjects matched according to age (18-40 years and 40-55 years) and with HIV positive subjects, vaccinated at J0 and followed over one year
  Interventions: Biological: Yellow fever vaccination (STAMARIL)

INTERVENTIONS:
Biological: Yellow fever vaccination (STAMARIL) — Yellow fever vaccination (STAMARIL)
Biological: Yellow fever vaccination (STAMARIL) — Yellow fever vaccination (STAMARIL)
  Arms: HIV negative subjects

SUMMARY:
Main objective :

To develop the tools for evaluation of humoral and cell-mediated immunity after Yellow Fever Vaccine (YFV) and compare virological and immune responses in HIV-positive and HIV-negative individuals who had not been given YFV before.

Secondary objectives :

* To develop and assess ELISPOT technology for yellow fever and to measure the response within 7, 14, 28, 90 and 365 days of administration of YFV in 30 HIV negative subjects and 40 HIV positive subjects (CD4 > 350/mm3 under Highly Active Antiretroviral Therapy (HAART) for at least one year, with a viral load < 50 copies/mL since at least 6 months) in terms of : (1) seroconversion by fluorescence, (2) cytotoxic response in ELISPOT, (3) neutralizing antibody levels in Plaque reduction neutralization test (PRNT:reference method) and a new pseudotype based method, (4) post-vaccination viremia and (5) diversity of viral quasi-species.
* To assess the impact of YFV on the T-lymphocyte response against HIV by ELISPOT and viral load.

DETAILED DESCRIPTION:
Method :

Clinical Trial Phase III, Multicentre protocol at Saint-Louis hospital, Bichat hospital and Cochin-Pasteur hospital, with CERVI, INSERM U 941 and SC10 collaboration.

Trial treatment : Yellow fever vaccination (STAMARIL)

Criterion :

Immuno-virologic: At J-7, J7, J28, M3 and M12 will be determined the levels of antibodies by fluorescence, at J0, J7, J28, M3 and M12 titles and neutralization with Prnt pseudotypes, the ELISPOT response anti-yellow fever, viremia with quantitative analysis and nucleotide sequences on phylogenetic strains of viremia. Titles and Amariles kinetics of viremia, neutralizing antibodies and ELISPOT will be considered as surrogate markers of response in terms of groups.

Clinical and biological tolerance: At all follows up will be measured the incidence of CDC classification events (for HIV+) and general and local reactions of degree ≥ 2 in the setting of the injection of STAMARIL®.

Schedule :

Date of first enrolment : third quarter 2011. Inclusion period : 18 months. For each subject, participation in this trial will be for 12 months.

ELIGIBILITY:
Group 1: Voluntary HIV positive subjects

Inclusion Criteria:

* Adults under HAART for at least one year (and stable on treatment for at least 3 months prior to enrolment)
* > 350 CD4/mm3 (with half of them a nadir < 200 CD4/mm3) and a viral load < 50 copies/mL for at least 6 months.
* Patients were HCV negative or non-replicative and treated for at least 2 years with normal ALT and negative HBs antigen.

Exclusion Criteria:

* Previous vaccination against yellow fever or yellow fever Fluorescence anti-IgG positive.
* Administration of immunoglobulins < 3 months or any vaccine <1 month.
* Pregnancy ongoing or planned during the study.
* Coinfection with HCV virus untreated.
* HBs Ag positive.
* Hypersensitivity reaction to eggs / chicken protein; hereditary fructose intolerance.
* Immunosuppression, whether congenital, idiopathic or as a result of corticosteroids systemically (at doses ≥ 20mg/d of prednisone), or due to radiation or antineoplastic older than 6 months.
* History of thymic dysfunction (including thymoma and thymectomy).
* For HIV + subjects: ART Celsentri or by other anti-CCR5.

Group 2: HIV negative subjects

Inclusion Criteria:

HIV and HCV negatives

Exclusion Criteria:

* Previous vaccination against yellow fever or yellow fever Fluorescence anti-IgG positive.
* Administration of immunoglobulins < 3 months or any vaccine <1 month.
* Other vaccinations should be deferred beyond M3.
* Pregnancy ongoing or planned during the study.
* Coinfection with HCV virus untreated.
* HBs Ag positive.
* Hypersensitivity reaction to eggs / chicken protein; hereditary fructose intolerance.
* Immunosuppression, whether congenital, idiopathic or as a result of corticosteroids systemically (at doses ≥ 20mg/d of prednisone), or due to radiation or antineoplastic older than 6 months.
* History of thymic dysfunction (including thymoma and thymectomy).
* For HIV + subjects: ART Celsentri or by other anti-CCR5, coinfection with HCV virus untreated

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2011-07; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Immuno-virologic criterion | DAY-7
  - At Day-7 will be determined the levels of antibodies by fluorescence.
Immuno-virologic criterion | Day 0
  At Day 0 will be determined titles and neutralization with Prnt pseudotypes, the ELISPOT response anti-yellow fever, viremia with quantitative analysis and nucleotide sequences on phylogenetic strains of viremia
Immuno-virologic criterion | Day 28
  At Day 28 will be determined titles and neutralization with Prnt pseudotypes, the ELISPOT response anti-yellow fever, viremia with quantitative analysis (if it's positive at day7) and nucleotide sequences on phylogenetic strains of viremia
Immuno-virologic criterion | Month 3
  At Month 3 will be determined fluorescence, PRNT and ELISPOT.
Immuno-virologic criterion | Month 12
  At Month 12 will be determined fluorescence, PRNT and ELISPOT.
Immuno-virologic criterion | Day 7
  At Day 7 will be determined titles and neutralization with Prnt pseudotypes, the ELISPOT response anti-yellow fever, viremia with quantitative analysis and nucleotide sequences on phylogenetic strains of viremia

SECONDARY OUTCOMES:
Clinical and biological tolerance | day -7
  At Day -7 will be determined the levels of antibodies by fluorescence
clinical and biological tolerance | day 0
  At Day 0: incidence of HIV+ event and general+local reactions of d°>2 after vaccination
clinical and biological tolerance | day 7
  At Day7: incidence of HIV+ event and general+local reactions of d°>2 after vaccination
clinical and biological tolerance | day 14
  At Day14:incidence of HIV+ event and general+local reactions of d°>2 after vaccination
clinical and biological tolerance | day 28
  At Day 28:incidence of HIV+ event and general+local reactions of d°>2 after vaccination
clinical and biological tolerance | month 3
  At Month3:incidence of HIV+ event and general+local reactions of d°>2 after vaccination
clinical and biological tolerance | month 12
  At Month 12:incidence of HIV+ event and general+local reactions of d°>2 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie COLIN de VERDIERE, Principal Investigator — Maladies Infectieuses St Louis Paris; Sophie MATHERON, Principal Investigator — Maladies Infectieuses et Tropicales Bichat Paris; Odile LAUNAY, Principal Investigator — CIC Cochin Paris
Locations (1):
- Voir Liste Des Centres, Paris, France

REFERENCES:
- [Derived] Colin de Verdiere N, Durier C, Samri A, Meiffredy V, Launay O, Matheron S, Mercier-Delarue S, Even S, Aboulker JP, Molina JM, Autran B, Simon F; ANRS EP46 NOVAA Group. Immunogenicity and safety of yellow fever vaccine in HIV-1-infected patients. AIDS. 2018 Oct 23;32(16):2291-2299. doi: 10.1097/QAD.0000000000001963. PMID 30096071
- See also: Related Info — http://anrs.fr